CLINICAL TRIAL: NCT05935072
Title: Nutritional Responses to Acute Exercise: Test of the Influence of the Nature of the Meal: EXHALIM Study
Brief Title: Nutritional Responses to Acute Exercise: Test of the Influence of the Nature of the Meal:
Acronym: EXHALIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2023 BOIRIE; 2023-A00687-38 (Other: ANSM)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Appetite Control; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rest with fixed meal (Experimental)
  Interventions: Behavioral: Exercice and meal
- rest with ad libitum meal (Experimental)
  Interventions: Behavioral: Exercice and meal
- Exercise with fixed meal (Experimental)
  Interventions: Behavioral: Exercice and meal
- Exercise with ad libitum meal (Experimental)
  Interventions: Behavioral: Exercice and meal

INTERVENTIONS:
Behavioral: Exercice and meal — The participants will carry out four experimental visits in a randomized order: CON_Calibré: control condition with a calibrated test meal; CON_AdLib: control condition with an ad libium test meal; EX_Calibré: exercise condition with a calibrated test meal; EX_AdLib: exercise condition with an ad libitm test meal. During each of the conditions, the participants will join the laboratory at 8:00 a.m. and will receive a calibrated breakfast. They will be asked at 11:00 a.m. either to rest in a semi-recumbent position for 30 minutes (CON conditions) or to perform a pedaling exercise on an ergocycle at 65% of their estimated aerobic capacity for 30 minutes. A test meal will be served to participants at 12:00 p.m., either ad libitum or calibrated. Appetite sensations will be assessed at regular intervals during each condition and their food reward preferences and ratio assessed 15 minutes before and 15 minutes after the test meals.

SUMMARY:
The management of body mass and energy balance requires a better understanding and mastery of the interactions between our daily activities, such as physical exercise, and the control of our food intake.

Over the past 15 years, many studies have focused on the potential effects of physical exercise on this satiety cascade and on subsequent food intake, in many populations. Thus, both in normal-weight subjects and in patients suffering from overweight and obesity, it has been shown that the performance of an acute exercise of moderate intensity promotes a transient anorectic effect, reducing feelings of hunger post -exercise, and can even induce a reduction in subsequent food intake. In healthy young adults, recent results show that high-intensity physical exercise can reduce feelings of hunger and increase the satietogenic effect of a meal compared to a control condition and low-intensity exercise. intensity. Nevertheless, it seems that the food reward (which refers to the notion of food reward) does not respond in the same way, the authors not observing any change in either liking or wanting, regardless of exercise intensity. Importantly, this literature uses ad libitum test meals, wishing to assess both satietogenic, hedonic and purely nutritional responses (assessing the amount of food intake). Nevertheless, these sensory and hedonic responses to food intake have recently been shown to be sensitive to the composition of the meal and its caloric quantity, which could induce a significant bias as to the conclusions on the effects of physical exercise. Indeed, the use of meals ad libitum, by definition, leads to caloric intake and different meal compositions. Thus, it is possible that the results obtained are strongly impacted by the nature of the test meal more than by the exercise itself. It therefore remains uncertain today to conclude as to the effects of physical exercise on the factors of the satietogenic cascade, since beyond physical exercise, the test meals compared are not identical. It therefore seems important today to develop a more coherent and adapted methodology, to better study the food and satietogenic responses to our daily activities.

In this context, the present project aims to compare the satietogenic response to a meal following acute exercise according to the nature of this meal (ad libitum versus calibrated) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 to 30 (limits inclusive),
* with a body mass index between 20 and 25 kg.m².
* Able to give informed consent to participate in research
* Person subject to a Social Security scheme

Exclusion Criteria:

* Medical or surgical history deemed by the investigator to be incompatible with the study.
* Presence of diabetes, and any other pathology limiting the application of one or the other strategy being tested.
* Subjects undergoing energy restriction or weight loss program through physical activity at the time of inclusion or during the last 6 months.
* Taking medications that may interfere with study results
* Claustrophobia
* Subjects with cardiovascular problems, here we are talking about subjects with a history of cardiovascular and/or neurovascular pathology, as well as subjects presenting cardiovascular and/or neurovascular risk factors (excluding obesity/ overweight).
* Student or professional in the field of dietetics and nutrition
* Surgical intervention in the previous 3 months.
* Person under guardianship / curatorship or safeguard of justice
* Participant refusal to participate Person in period of exclusion from another study
* Tobacco use
* Alcohol consumption (more than 5 drinks per week).
* Special diet.
* Participation in regular and intense physical and sports activities (more than 90 minutes per week).
* Person refusing to be registered on the National File of Healthy Volunteers of the Ministry of Health,
* Subject in a period of exclusion from a previous study or having received a total amount of compensation greater than 6000 euros over the 12 months preceding the start of the trial (after verification in the Biomedical Research Volunteers File).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Satiety Quotient | During every experimental sessions, right after the lunch
  Ratio between the energy content of the meal and the self-reported appetite feelings

SECONDARY OUTCOMES:
Food reward | During every experimental sessions,15 minutes before and 15 minutes after the lunch
  The liking and wanting for food items using a computerized questionnaire
Ad libitum food intake | During every experimental sessions at diner
  energy ingested at a diner buffet meal

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France